CLINICAL TRIAL: NCT04708379
Title: Lifestyle Interventions for Overweight Adults With Severe Mental Illness in Shenzhen, China
Brief Title: Lifestyle Interventions for Overweight Adults With Mental Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wuhan University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Qiqiang He, Professor, Wuhan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pingshan Mental Health Study
Record Dates: First submitted 2021-01-03; First posted 2021-01-13 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Mental Health Disorder
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Nutrition education and physical activity education.
  Interventions: Behavioral: Lifestyle intervention
- Control group (No Intervention): No specific intervention.

INTERVENTIONS:
Behavioral: Lifestyle intervention — Nutrition and physical activity education.
  Arms: Intervention group

SUMMARY:
The purpose of this study is to examine the lifestyle intervention on life quality and mental health among overweight adults with severe mental illness in Shenzhen, China. A total of 210 overweight adults with severe mental illness will be randomly allocated to intervention group and control group. Participants in the intervention groups will receive a 10-month lifestyle intervention while the control group will be waitlisted. A group of investigators will measure the anthropocentric indicators, blood pressure, lifestyle, life quality, and mental health for all participants.

DETAILED DESCRIPTION:
Previous studies suggest that overweight is an important risk factor for life quality and mental health among patients with severe mental illness. Findings on Chinese adults regarding this issue are limited. Thus, we aim to assess the lifestyle intervention on life quality and mental health among overweight adults with severe mental illness in Shenzhen, China.

A total of 210 overweight adults with severe mental illness will be randomly allocated to two groups. Participants in the intervention groups will receive a 10-month lifestyle intervention while the control group will be waitlisted.

In the intervention group, participants will receive lifestyle education delivered by trained staffs from Wuhan university. The main objective of the lifestyle education is to raise participants' awareness regarding the health complications related to obesity and subsequently to promote weight loss through behavioural modifications. Participants will be advised to reduce energy intake by having three main meals and avoiding snacks; limiting intake of sugary food and beverages as well as fried and fatty foods; increasing intake of fruits and vegetables, etc. They will be asked to increase physical activity, aiming for a minimum 150 min of moderate-intensity exercise per week and/or 10,000 steps per day.

Outcome measurement include height, weight, blood pressure, dietary habits, sleep, physical activity, life quality, and mental health that will be measured by a group of trained investigator for all participants.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years
* With severe mental illness
* BMI>=24.0
* Live in this district for 1 year at least.

Exclusion Criteria:

* Disability
* Refuse to participate
* Pregnant woman
* Severe chronic diseases, such as cancer.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
BMI | 12 weeks
  Participants' height (in meters) and weight (in kilograms) will be measured by a group of investigators. weight and height will be combined to report BMI in kg/m^2.

SECONDARY OUTCOMES:
Life quality | 12 weeks
  Life quality will be investigated by the short form version of the quality of life enjoyment and satisfaction questionnaire (Q-LES-Q-SF). Each item uses a 5-point scale ranging from 1 (very poor) to 5 (very good). A total score is derived from 14 items with a maximum score of 70 and with higher scores indicating greater life satisfaction and enjoyment.
Depression | 12 weeks
  Depression will be assessed by Center for Epidemiological Studies Depression Scale (CES-D). This is a 20-item measure that asks participants to rate how often over the past week they experienced symptoms associated with depression. Response options range from 0 to 3 for each item. Scores range from 0 to 60, with high scores indicating greater depressive symptoms.
Social support | 12 weeks
  Social support will be assessed by Perceived social support scale(PSSS). The scale consists of 12 items, including family support, friend support and other support. The higher the score of Liker-7 points, the higher the level of social support perceived by the individual.

OTHER OUTCOMES:
BP | 12 weeks
  Blood pressure (measured by a group of investigators)
Sleep | 12 weeks
  Sleep status will be assessed by Pittsburgh Sleep Quality Index (PSQI). The PSQI is a self-report questionnaire consisting of 19 items and five additional questions. The 19 items are combined to form seven sleep quality component scores. Each component score can range from 0 to 3. The seven component scores are summed to yield a global PSQI score ranging from 0 to 21, with higher scores indicate poorer sleep quality.
Physical activity | 12 weeks
  Physical activity will be assessed by International Physical Activity Questionnaire (IPAQ). This IPAQ consists of seven questions assessing the frequency and duration of participation in vigorous, moderate-intensity, and walking activity as well as the time spent sitting during a weekday. The sum of the three activity scores gives an indicator of total physical activity.
Diet | 12 weeks
  Participants self-report their dietary intake including rice, meat, milk, fruits, vegetable, etc using a short food frequency questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Qiqiang He, PhD, Principal Investigator — Wuhan University
Locations (1):
- Pingshan CDC, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No